CLINICAL TRIAL: NCT04024215
Title: Role of Intravascular Ultrasound(IVUS) in Management of Acute and Chronic Iliocaval Obstruction
Brief Title: Role of IVUS in Management of Iliocaval Obstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Hamdi Ali Abdel-kader, Principal Investigator, Assiut University
Other Study IDs: IVUS in iliocaval obstruction
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Iliocaval Compression Syndrome
Keywords: intravascular ultrasound
MeSH Terms: conditions — May-Thurner Syndrome | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intravascular ultrasound — IVUS creates axial images perpendicular to the long axis of the catheter by transmitting sound waves covering 360 degrees around the tip of the catheter, which is delivered into the lumen of the vessel over a guidewire.

SUMMARY:
To assess the role of IVUS in

1. Providing diagnostic important data as: luminal diameters, cross-sectional area, assessment of potential thrombus volume which enables optimal choice of appropriate angioplasty technique, endovascular device guidance, and their impact on procedural technical success and patency rates.
2. comparing diagnostic accuracy of intravascular ultrasound (IVUS) with multiplanar venography and CT venography for iliocaval obstruction.

DETAILED DESCRIPTION:
Acute and chronic venous disorders of the lower extremities affect millions of people and cause substantial disability. Surgeons and pathologists identified the presence of 'spur-like' abnormalities of the left common iliac vein, these abnormalities were hypothesized to result from compression and/or irritation from the adjacent crossing right common iliac artery. In the 1990s, physicians, starting to perform catheter-directed thrombolysis to treat extensive deep vein thrombosis (DVT), observed that about 50% of patients had an iliac vein stenosis.Treatment is aimed at ameliorating the symptoms and, whenever possible, at correcting the underlying abnormality. Graduated compression is the cornerstone of modern therapy. Deep system disease is often refractory to treatment, but superficial system disease can usually be treated by ablating the refluxing vessels. Effective venous return from the lower extremities requires the interaction of the heart, a pressure gradient, the peripheral muscle pumps of the leg, and competent venous valves. In the absence of pathology, this system functions to reduce venous pressure from approximately 100 mm Hg to a mean of 22 mm Hg within a few steps.

Nonthrombotic venous compression patients with left common iliac vein compression can present in the 2nd or 3rd decade of life and are more common in women. Patients can have limb pain, limb swelling, ipsilateral chronic venous insufficiency, lipodermatosclerosis, recurrent superficial venous thrombophlebitis, and venous claudication.

Thrombotic iliofemoral venous compression with a predisposing anatomic configuration with a prothrombotic physiological state can present with acute pain and swelling of the left lower extremity consistent with an acute iliofemoral DVT mostly phlegmasia cerulea dolens . In the acute phase, patients with a patent foramen ovale can also present with a pulmonary embolism, cryptogenic stroke, with or without pulmonary embolism, or systemic arterial embolism.

The abnormalities in venous physiology associated with chronic venous disease, and their quantification by diagnostic tests, are also considerably more complex than for PAD. With CVD one must gauge the effects of obstruction and/or reflux in a vascular bed uniquely designed to return venous blood to the heart against gravity with the aid of a peripheral muscle pump and in phase with respiratory mechanics.

Duplex ultrasound (DUS) is initial diagnostic test. The criteria include: poststenotic turbulence, as indicated by a mosaic velocity profile, abnormal Doppler signal at the area of stenosis, continuous flow with the Valsalva maneuver, and sluggish with no spontaneous flow and poor augmentation and no respiratory phasicity. But there is limitations as obesity ,casts, dressings, open wounds, Patients with severe edema/swelling and limited patient mobility.

Cross-sectional imaging includes computed tomographic venography (CTV) with venous phase contrast or magnetic resonance venography (MRV).

Catheter-based phlebography traditionally is considered to be the most definitive technique for the evaluation of venous obstruction, supplemented with direct pressure measurements across an area of perceived stenosis in order to determine whether a pressure gradient exists.

Intravascular ultrasound (IVUS) uses a catheter-based ultrasound probe that enables high-resolution evaluation of the vein wall and internal venous architecture in 360. IVUS is more sensitive than phlebography for the detection and characterization of iliac vein pathology. This would be expected since IVUS gives a 360 image versus a single plane image shown by standard phlebograms. Intravascular ultrasound also identifies intraluminal trabeculations, septations, webs, and wall thickening, which can be minimized or missed on standard phlebography, plus reduced radiation exposure in contrast to other modalities.

IVUS is better in evaluating lesion morphology, accurate assessment of luminal dimensions, transmural lesion characteristics. Delineation by IVUS of the spatial distribution of the lesion in a concentric or eccentric pattern and the presence of a soft (fibrous) or hard (calcified) plaque may influence the choice of endovascular therapy as well as predict the risk of immediate or late complications (ie, perforation, thrombosis, restenosis). Evaluation of lesion volume before and after the procedure by IVUS provides a quantitative method to estimate the amount of lesion debulking or displacement and a reference point from which to assess the lesion recurrence/restenosis. IVUS also fulfills many of the necessary requirements of a guidance system for endovascular procedures, namely precise delivery and positioning of stents within target lesions. IVUS is particularly helpful in assessing the relationship of the ostia of branch vessels to the lesion that can be used as landmarks during procedures.

ELIGIBILITY:
Inclusion Criteria:

* 1-acute iliocaval obstruction 2-chronic iliocaval obstruction with CEAP clinical class 3-6 3- acute on top of chronic iliocaval obstruction with CEAP clinical class 3-6 4-symptomatic acute femoro-iliocaval occlusion who underwent successful thrombolysis

Exclusion Criteria:

1 - concomitant peripheral arterial disease in the affected limb. 2-life expectancy less than 5 years. 3- pregnancy 4- malignancy 5-raised renal chemistry 6-pelvic fibrosis 7- contraindication to anti-coagulation therapy. 8-congenital venous malformations 9-Not providing informed consent 10-Any concurrent disease as heart failure

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: subjects with with acute or chronic iliocaval obstruction CEAP classification 3-6.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage diameter change in iliocaval segment | baseline
  Compare the percentage diameter reduction measured by intravascular ultrasound (IVUS) and venography and interventional venogram
Percentage area change in iliocaval segment | baseline
  Compare the percentage area reduction measured by IVUS and the calculated percentage area reduction measured by venography and interventional venogram
technical success of the preformed procedure of endovascular intervention | baseline
  patency of the treated vessel segment with\20 % residual stenosis and without dissection or extravasation.

SECONDARY OUTCOMES:
Primary Patency of the performed procedure | baseline
  uninterrupted vessel patency with no procedure performed on the treated segment.
Secondary Patency of the performed procedure | baseline
  whenever maintenance of patency required secondary intervention at the target lesion.
Assisted Primary Patency of the performed procedure | baseline
  cases in which a revision of the revascularization method is applied before vessel occlusion occurs as prophylactic interventions.

CONTACTS AND LOCATIONS:
Overall Officials: moustafa saad khalil, professor, Study Director — Assiut University; hesham aboelyoun, lecturer, Study Chair — Assiut University; ahmed hassan bakr, A.professor, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renner R, Gebhardt C, Simon JC, Seikowski K. Changes in quality of life for patients with chronic venous insufficiency, present or healed leg ulcers. J Dtsch Dermatol Ges. 2009 Nov;7(11):953-61. doi: 10.1111/j.1610-0387.2009.07082.x. English, German. PMID 19386020
- [Background] Labropoulos N, Borge M, Pierce K, Pappas PJ. Criteria for defining significant central vein stenosis with duplex ultrasound. J Vasc Surg. 2007 Jul;46(1):101-7. doi: 10.1016/j.jvs.2007.02.062. Epub 2007 May 30. PMID 17540535
- [Background] Forauer AR, Gemmete JJ, Dasika NL, Cho KJ, Williams DM. Intravascular ultrasound in the diagnosis and treatment of iliac vein compression (May-Thurner) syndrome. J Vasc Interv Radiol. 2002 May;13(5):523-7. doi: 10.1016/s1051-0443(07)61535-8. PMID 11997362
- [Background] Neglen P, Raju S. Intravascular ultrasound scan evaluation of the obstructed vein. J Vasc Surg. 2002 Apr;35(4):694-700. doi: 10.1067/mva.2002.121127. PMID 11932665
- [Background] Vedantham S, Grassi CJ, Ferral H, Patel NH, Thorpe PE, Antonacci VP, Janne d'Othee BM, Hofmann LV, Cardella JF, Kundu S, Lewis CA, Schwartzberg MS, Min RJ, Sacks D; Technology Assessment Committee of the Society of Interventional Radiology. Reporting standards for endovascular treatment of lower extremity deep vein thrombosis. J Vasc Interv Radiol. 2009 Jul;20(7 Suppl):S391-408. doi: 10.1016/j.jvir.2009.04.034. No abstract available. PMID 19560027
- [Result] Buckley CJ, Arko FR, Lee S, Mettauer M, Little D, Atkins M, Manning LG, Patterson DE. Intravascular ultrasound scanning improves long-term patency of iliac lesions treated with balloon angioplasty and primary stenting. J Vasc Surg. 2002 Feb;35(2):316-23. doi: 10.1067/mva.2002.119755. PMID 11854730
- See also: CIRSE Standards of Practice Guidelines on Iliocaval Stenting — http://link.springer.com/article/10.1007%2Fs00270-014-0875-4